CLINICAL TRIAL: NCT05629767
Title: Tracking Lipid-Lowering Therapy Over One Year in Middle Eastern Patients With ASCVD. The Jordan LLA Tracking Study
Brief Title: Tracking of Lipid Lowering Therapy in Jordan
Acronym: JoLLA
Status: Terminated | Type: Observational
Why Stopped: Inadequate enrolling numbers of patients
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: JCCG.JoLLA.10.2022
Record Dates: First submitted 2022-10-29; First posted 2022-11-29 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Dyslipidemias; Atherosclerotic Cardiovascular Disease
Keywords: Low-density lipoprotein cholesterol (LDL-C), Target levels
MeSH Terms: conditions — Dyslipidemias; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ASCVD: Patients with ASCVD on statins and LDL-C more than 70 mg/dl

SUMMARY:
The present study aims to examine the clinical practice of modifying the dose of lipid-lowering therapy in patients with atherosclerotic cardiovascular disease (ASCVD), who have LDL-C > 70 mg/dl despite statin treatment.

DETAILED DESCRIPTION:
ASCVD is the leading cause of morbidity and mortality worldwide, in the Middle East and in Jordan. One of the major risk factors that contribute to the development and progression of ASCAD is dyslipidemia. A large number of clinical trials have reported the benefits of lowering LDL-C, in reducing the mortality rate among ASCAD patients.

The 2019 ACC/AHA blood cholesterol treatment guideline to reduce atherosclerotic cardiovascular risk in adults has expanded the role of LDL-C targets and reiterated the importance of achieving an LDL-C level of 70 mg/dl or less for patients who have ASCVD.

Patients on statins and other lipid-lowering therapy in Jordan have not been tracked in the past for the potential of up escalating the lipid-lowering therapy to reach the LDL-C target.

The investigation will enroll patients with ASCVD who have LAL-C >70 mg/dl on lipid-lowering therapy and follow them for 12 months to examine the treating physicians' action in up-titrating the lipid-lowering therapy dose(s) and the frequency of measuring serum lipids during the study period.

ELIGIBILITY:
Inclusion criteria

1. Adults aged 18 years or old.
2. Presence of atherosclerotic cardiovascular disease on lipid-lowering therapy.
3. LDL-C > 70mg/dl.
4. Willingness to sign an informed consent.

Exclusion criteria

1. Life-threatening disease with limited survival.
2. Unwillingness to sign an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll adults aged 18 years or old with a diagnosis of atherosclerotic cardiovascular disease on lipid-lowering therapy (statins and non-statins) and an LDL-C > 70mg/dl. and follow them up for 12 months to evaluate the up-titrating of the lipid-lowering therapy and the frequency of repeating the lipid measurement.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-12-11 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Achieving a target LDL-C bloob level of 70 mg/dl or less | 12 months
  At 1 year of follow up, all participants will have their blood lipid profile measured to examine the frequency of attaining an LDL-C level of 70 mg/dl or less
Modifying the dose and class of lipid-lowering therapy | 12 months
  Up titrating the dose of the same lipid-lowering agent or adding new agent during the study period of 12 months. Agents available include statins, ezetimibe and PCSK9 inhibitors.
Clinical cardiovascular events | 12 months
  The study will study the frequency of incident acute cardiovascular the participating individuals experienced. Such events include cardiovascular death, acute coronary syndrome, stroke, lower extremity acute arterial insufficiency, and arterial revascularization procedure (coronary and other arterial beds).

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Hammoudeh, MD FACC, Principal Investigator — Istishari Hospital, Amman, Jordan
Locations (2):
- Jordan (2):
  - Istishari Hospital, Amman
  - Abdali Hospital, Amman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shi A, Tao Z, Wei P, Zhao J. Epidemiological aspects of heart diseases. Exp Ther Med. 2016 Sep;12(3):1645-1650. doi: 10.3892/etm.2016.3541. Epub 2016 Jul 26. PMID 27602082
- [Result] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2889-934. doi: 10.1016/j.jacc.2013.11.002. Epub 2013 Nov 12. No abstract available. PMID 24239923
- [Result] Wilson PWF, Polonsky TS, Miedema MD, Khera A, Kosinski AS, Kuvin JT. Systematic Review for the 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Jun 25;73(24):3210-3227. doi: 10.1016/j.jacc.2018.11.004. Epub 2018 Nov 10. PMID 30423394
- [Result] Bloom BS. Effects of continuing medical education on improving physician clinical care and patient health: a review of systematic reviews. Int J Technol Assess Health Care. 2005 Summer;21(3):380-5. doi: 10.1017/s026646230505049x. PMID 16110718
- [Result] Santi RL, Martinez F, Baranchuk A, Liprandi AS, Piskorz D, Lorenzatti A, Santi MPL, Kaski JC. Management of Dyslipidaemia in Real-world Clinical Practice: Rationale and Design of the VIPFARMA ISCP Project. Eur Cardiol. 2021 Apr 27;16:e16. doi: 10.15420/ecr.2020.42. eCollection 2021 Feb. PMID 33995586

DOCUMENTS (1):
  • Study Protocol (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT05629767/Prot_000.pdf